CLINICAL TRIAL: NCT01669798
Title: Phase II Evaluation of BIBF 1120 in the Treatment of Bevacizumab-Resistant, Persistent, or Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma
Brief Title: BIBF 1120 in Bevacizumab Resistant, Persistent, or Recurrent Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AA Secord (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, AA Secord, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00033060
Record Dates: First submitted 2012-07-10; First posted 2012-08-21 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
Keywords: Recurrent epithelial ovarian carcinoma; Persistent epithelial ovarian carcinoma; Bevacizumab resistant epithelial ovarian carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- BIBF 1120 (Experimental): BIBF 1120 will be administered at a daily oral dose of 200 mg BID until disease progression or adverse effects prohibit further therapy.
  Interventions: Drug: BIBF 1120

INTERVENTIONS:
Drug: BIBF 1120 — PO 200mg BID
  Other Names: Vargatef™; Nintedanib

SUMMARY:
The main purpose of this study is to see if BIBF 1120 can increase the number of women with bevacizumab resistant, persistent, or recurrent epithelial ovarian cancer who do not progress for at least six months.

DETAILED DESCRIPTION:
Ovarian cancer patients with platinum-resistant and refractory disease have the lowest response rates to relapse chemotherapy: various chemotherapeutic agents, such as paclitaxel, liposomal doxorubicin, topotecan, docetaxel, platinum, etoposide, ifosfamide, gemcitabine, and vinorelbine are available but result in response rates of 7-40%. Unfortunately, relapse therapy is not curative and treatment is only palliative. Recently two phase II trials demonstrated that anti-angiogenic therapy with bevacizumab alone or in combination with chemotherapy in women with recurrent disease had response rates ranging from 16-24% with an acceptable toxicity profile. However, resistance can develop to VEGF inhibition. Therefore other novel anti-angiogenic agents, such as BIBF 1120, should be evaluated in the treatment of ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma w/ histologic documentation of the original primary tumor via the pathology report:

  * serious, endometrioid, mucinous, or clear cell adenocarcinoma
  * undifferentiated, mixed epithelial or transitional cell carcinoma
  * Brenner's Tumor
  * adenocarcinoma NOS
* Had treatment-free interval following response to bevacizumab (CR, PR, or SD) of < 6 months, or have progressed during treatment w/ a bevacizumab-containing therapy
* Measurable or detectable disease. Measurable is defined by RECIST 1.1. Each lesion must be ≥ 10 mm when measured by CT, MRI or caliper measurement by clinical exam; or ≥ 20 mm when measured by chest x-ray. Lymph nodes must be > 15 mm in short axis when measured by CT or MRI. Detectable defined as no measurable disease but either ascities/pleural effusion or solid/cystic abnormalities that don't meet RECIST 1.1 - both within the setting of CA125 >2xULN
* Those with measurable disease must have at least one "target lesion" to assess response as defined by RECIST 1.1. Tumors in a previously irradiated field will be designated as "non-target" lesions
* Must have a ECOG Performance Status of 0 or 1
* Free of active infection requiring antibiotics. Exception: uncomplicated UTI
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy

  * Hormonal therapy directed at the malignant tumor must be d/c at least a week prior to registration. Hormone replacement therapy is permitted
  * Other prior therapy directed at malignant tumor, including immunologic agents, must be d/c at least 3 weeks prior to registration; 4 weeks if prior therapy was w/ bevacizumab
* Prior therapy

  * must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound. This initial treatment may have included intraperitoneal therapy, high-dose therapy, consolidation, non-cytotoxic agents or extended therapy administered after surgical or non-surgical assessment.
  * Allowed, to receive, but not required to receive, 2 additional cytotoxic regimens for management of recurrent or persistent disease according to the following:

    * Patients who have received only one prior cytotoxic regimen (platinum-based regimen for management of primary disease), must have a platinum-free interval of less than 12 months, or have progressed during platinum-based therapy, or have persistent disease after a platinum-based therapy.
    * Patients must NOT have received any non-cytotoxic therapy for management of recurrent or persistent disease other than bevacizumab. Patients are allowed to receive, but are not required to receive, biologic (non-cytotoxic) therapy as part of their primary treatment regimen.
* Must have adequate:

  * Bone marrow function: Absolute neutrophil count (ANC) ≥ 1,500/mcl, equivalent to (CTCAE v4.0) grade 1. Platelets ≥ 100,000/mcl. Hemoglobin (Hb) ≥ 9.0 g/dL
  * Renal function: creatinine ≤ 1.5 x upper limit of normal (ULN)
  * Hepatic function: Bilirubin should be w/in normal limits (CTCAE v4.0, grade 1). ALT/AST, should be ≤ 1.5 x ULN (CTCAE v4.0, grade 1). For patients w/ liver metastases, ALT/AST should be ≤ 2.5 x ULN; Alkaline phosphatase should be ≤ 2.5 x ULN (CTCAE v4.0, grade 1)
  * Neurologic function: Neuropathy ≤ CTCAE v4.0, grade 1
* Blood coagulation parameters: PT w/ international normalized ratio (INR) < 1.5 x ULN & a PTT < 1.5 x ULN (or an in-range PTT if on a stable dose of therapeutic heparin). Low molecular weight heparin (enoxaparin or alternative anticoagulants (other than warfarin)) are acceptable.
* Signed informed consent & authorization permitting release of personal health information
* Negative serum pregnancy test if of childbearing potential prior to study entry & use of effective form of contraception until 3 months after receiving last drug treatment
* Patients may have undergone a major or minor surgical procedure as long as:

  * > 28 days prior to the first date of study therapy
  * Core biopsy or IV Port placement greater than 7 days prior to the first date of study therapy

Exclusion Criteria:

* Previous treatment w/ BIBF 1120.
* Pregnant or breastfeeding.
* Received radiation to more than 25% of marrow-bearing areas
* History of other invasive malignancies, w/ the exception of non-melanoma skin cancer, if there is any evidence of other malignancy being present w/in the last five years.
* Received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for treatment of ovarian, fallopian tube, or primary peritoneal cancer w/in the last 5 years.
* Prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer or localized breast cancer w/in the last 5 years.
* A history of abdominal or tracheal-esophageal fistula, or gastrointestinal perforation
* A history of intra-abdominal abcess w/in 6 months of enrollment
* Serious, uncontrolled, concomitant disorder(s) such as diabetes mellitus
* Patients w/ clinically significant cardiovascular disease including: uncontrolled hypertension: systolic > 150 mm Hg/diastolic > 90 mm Hg; unstable angina or who have had a myocardial infarction w/in the past six months prior to registration; congestive heart failure; cardiac arrhythmia requiring medication (doesn't include asymptomatic atrial fibrillation); grade 2 or greater peripheral vascular disease (at least brief (<24 hours) episodes of ischemia managed non-surgically & w/o permanent deficit.
* Serious non-healing wound, ulcer, or bone factor.

  o Granulating incisions healing by secondary intention w/ no evidence of fascial dehiscence or infection ARE eligible but require weekly wound examinations.
* Active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder, coagulopathy, or tumor involving major vessels.
* History/evidence upon physical examination of CNS disease, including primary brain tumor, seizures not controlled w/ standard medical therapy, any brain metastases, CVA, TIA, or subarachnoid hemorrhage w/in 6 months of the first date of treatment on this study.
* Central pulmonary metastases/recent hemoptysis (≥1/2 tsp of red blood) w/in 28 days of registration.

  * Clinically significant proteinuria (i.e. >Grade 1) or UPC ratio above 1.0
  * Suspicion of transmural tumor bowel involvement based on the investigator's discretion.
* Clinical symptoms/signs of gastrointestinal obstruction & require IV hydration &/or nutrition.
* Patients taking warfarin are not eligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-02; Primary Completion 2017-09-10 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angeles A Secord, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Duke Cancer Institute, Durham, North Carolina
  - University of Virginia, Charlottesville, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from February of 2013 to July of 2017 at three cancer clinics in North Carolina and Virginia.
Period: Overall Study
Arm/Group | BIBF 1120
Started | 32
Completed | 27
Not Completed | 5
Not completed — Physician Decision | 5

BASELINE CHARACTERISTICS:
Arm/Group | BIBF 1120
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 24
  More than one race | 0
  Unknown or Not Reported | 1
Primary site of tumor [Count of Participants; unit: Participants]
  Ovary | 26
  Peritoneum | 1
Histologic tumor type [Count of Participants; unit: Participants]
  Adenocarcinoma, Unspecified | 1
  Clear Cell Carcinoma | 1
  Other: Poorly Differentiated Adenocarcinoma | 1
  Serous Adenocarcinoma | 24
Platinum based treatment resistant/sensitive [Count of Participants; unit: Participants]
  Platinum Resistant | 22
  Platinum Sensitive | 5
Antecedent Bevacizumab (bev) therapy prior to starting trial [Count of Participants; unit: Participants]
  Front-line chemo with bev, plus bev maintenance | 9
  Front-line chemo with bev, without bev maintenance | 2
  Second-line chemo with bev, plus bev maintenance | 5
  Secon-line chemo with bev, without bev maintenance | 4
  Second line single agent bevacizumab | 6
  Third-line chemotherapy plus bevacizumab | 1
Number of prior therapy regimens [Count of Participants; unit: Participants]
  One prior regimen | 8
  Two prior regimens | 10
  Three prior regimens | 7
  Four prior regimens | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Survive Progression-free
Description: Measure of Progression Free Survival (PFS) by the percentage of patients who survive progression-free for at least 6 months after initiating study therapy in patients with bevacizumab-resistant, persistent or recurrent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.
Time Frame: 6 months
Population: The analysis was to be based on 27 evaluable patients for the first stage. Subjects were considered evaluable if they completed at least one cycle of study drug. Of the 27 subjects, one was not considered evaluable because they did not receive a full cycle.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIBF 1120
Number analyzed (Participants) | 26
percentage of participants | 11.5 [2.5 to 30.2]

2. Secondary Outcome: Objective Tumor Response Via RECIST (Response Evaluation Criteria in Solid Tumors) 1.1
Description: Evaluating the percentage of patients who have objective tumor response (complete or partial) based on RECIST 1.1 criteria.
Time Frame: 1 year
Population: Responders are those who achieved a partial response (PR). No subjects achieved a complete response (CR).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BIBF 1120
Number analyzed (Participants) | 27
percentage of participants | 7.4 [0.9 to 24.3]

3. Secondary Outcome: Duration of Progression-Free Survival
Description: The duration of progression-free survival and overall survival measured in months; Progression-Free Survival (PFS) is defined as the duration of time from study entry to time of progression or death, whichever occurs first.
Time Frame: Through study completion, on average 2 years
Population: Analysis stratified results between PFS (Progression Free Survival) and OS (Overall Survival). Confidence interval and results based on Kaplan Meier Estimates.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | BIBF 1120
Number analyzed (Participants) | 27
Months
  Progression Free Survival (PFS) | 1.8 [1.6 to 3.5]
  Overall Survival (OS) | 16 [8 to 25]

4. Secondary Outcome: Objective Tumor Response Based on GCIG CA-125 Criteria
Description: The proportion of patients who have objective tumor response (complete or partial) based on Gynaecologic Cancer InterGroup(GCIG) CA-125 criteria which is: "A response according to CA 125 has occurred if there is at least a 50% reduction in CA 125 levels from a pretreatment sample. The response must be confirmed and maintained for at least 28 days.".
Time Frame: 1 year
Population: Twenty five subjects were analyzed based on the Gynaecologic Cancer Intergroup response CA125 response criteria. Two subjects data were unavailable.
Measure: Count of Participants; unit: Participants
Arm/Group | BIBF 1120
Number analyzed (Participants) | 25
Participants | 0

5. Secondary Outcome: Adverse Event Frequency and Severity
Description: To determine frequency and severity of adverse events as assessed using NCI Common Toxicity Criteria version 4.
Time Frame: 1 year
Population: All adverse events considered possible, probably, or definitely related to study drug. Reported regardless of severity.
Measure: Count of Participants; unit: Participants
Arm/Group | BIBF 1120
Number analyzed (Participants) | 27
Participants
  Anemia | 2
  Sinus tachycardia | 1
  Tinnitus | 1
  Abdominal pain | 7
  Bloating | 3
  Diarrhea | 17
  Dry mouth | 1
  Constipation | 4
  Dyspepsia | 1
  Gastroesophageal reflux disease | 1
  Nausea | 17
  Vomiting | 13
  Chills | 1
  Edema limbs | 3
  Fatigue | 14
  Non-cardiac chest pain | 1
  Alanine aminotransferase increased | 10
  Alkaline phosphatase increased | 8
  Aspartate aminotransferase increased | 12
  Creatinine increased | 1
  Neutrophil count decreased | 1
  Platelet count decreased | 2
  Weight loss | 3
  Anorexia | 4
  Hypoalbuminemia | 2
  Hypocalcemia | 1
  Hypomagnesemia | 4
  Hyponatremia | 4
  Arthralgia | 4
  Arthritis | 1
  Back Pain | 2
  Bone pain | 1
  Pain in extremity | 1
  Dysgeusia | 2
  Headache | 8
  Hematuria | 1
  Proteinuria | 4
  Urinary incontinence | 1
  Vaginal dryness | 1
  Vaginal pain | 1
  Atelectasis | 1
  Dyspnea | 2
  Pleural effusion | 1
  Wheezing | 1
  Rash maculo-papular | 1
  Hypertension | 4
  Intermittent leg cramps | 1
  Bilateral neuropathy, hands and feet | 1

6. Other Pre Specified Outcome: Concentration of Select Growth Factors Reported Measured in Picograms Per Milliliter as a Function of Treatment Response
Description: Correlating baseline and on treatment levels of additional growth factors measured in picograms per milliliter that may be co- or counter- regulated with VEGF with response to treatment
Time Frame: 1 year
Population: Biomarker levels measured and stratified into two groups: those who experienced either Partial Response (PR) or Stable Disease (SD); and those who experienced Progressive Disease (PD). Data was not collected for one subject.
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter
Arm/Group | BIBF 1120
Number analyzed (Participants) | 26
picograms per milliliter
  CD73: Partial Response or Stable Disease: number analyzed (Participants) | 11
  CD73: Partial Response or Stable Disease | 3.0 [1.8 to 3.4]
  CD73: Progressive Disease: number analyzed (Participants) | 15
  CD73: Progressive Disease | 3.8 [2.6 to 5.0]
  HGF: Partial Response or Stable Disease: number analyzed (Participants) | 11
  HGF: Partial Response or Stable Disease | 130.1 [78.3 to 188.2]
  HGF: Progressive Disease: number analyzed (Participants) | 15
  HGF: Progressive Disease | 191.0 [72.1 to 517.4]
  IL-6: Partial Response or Stable Disease: number analyzed (Participants) | 11
  IL-6: Partial Response or Stable Disease | 18.2 [8.9 to 28.5]
  IL-6: Progressive Disease: number analyzed (Participants) | 15
  IL-6: Progressive Disease | 32.6 [16.5 to 50.5]
  PDGF-AA: Partial Response or Stable Disease: number analyzed (Participants) | 11
  PDGF-AA: Partial Response or Stable Disease | 89.5 [27.7 to 347.4]
  PDGF-AA: Progressive Disease: number analyzed (Participants) | 15
  PDGF-AA: Progressive Disease | 233.9 [47.1 to 419.6]
  PDGF-BB: Partial Response or Stable Disease: number analyzed (Participants) | 11
  PDGF-BB: Partial Response or Stable Disease | 184.7 [26.7 to 325.6]
  PDGF-BB (pg/ml): PD: number analyzed (Participants) | 15
  PDGF-BB (pg/ml): PD | 396.4 [91.1 to 769.2]
  PIGF: Partial Response or Stable Disease: number analyzed (Participants) | 11
  PIGF: Partial Response or Stable Disease | 23.4 [21.5 to 27.9]
  PIGF: Progressive Disease: number analyzed (Participants) | 15
  PIGF: Progressive Disease | 24.3 [14.2 to 30.5]
  SDF-1: Partial Response or Stable Disease: number analyzed (Participants) | 11
  SDF-1: Partial Response or Stable Disease | 1968.6 [1453.7 to 3021.0]
  SDF-1: Progressive Disease: number analyzed (Participants) | 15
  SDF-1: Progressive Disease | 2121.9 [1199.4 to 3360.0]
  TGFBeta-R3: Partial Respone or Stable Disease: number analyzed (Participants) | 11
  TGFBeta-R3: Partial Respone or Stable Disease | 50.6 [32.8 to 71.0]
  TGFBeta-R3: Progressive Disease: number analyzed (Participants) | 15
  TGFBeta-R3: Progressive Disease | 52.5 [45.4 to 57.3]
  Ang2: Partial Response or Stable Disease: number analyzed (Participants) | 11
  Ang2: Partial Response or Stable Disease | 261.1 [141.6 to 456.1]
  Ang2: Progressive Disease: number analyzed (Participants) | 15
  Ang2: Progressive Disease | 189.5 [146.7 to 222.5]
  BMP-9: Partial Response or Stable Disease: number analyzed (Participants) | 11
  BMP-9: Partial Response or Stable Disease | 47.0 [39.0 to 62.7]
  BMP-9: Progressive Disease: number analyzed (Participants) | 15
  BMP-9: Progressive Disease | 45.9 [36.2 to 48.3]

7. Other Pre Specified Outcome: Coagulation and Endothelial Cell Activation Markers
Description: To measure baseline and on treatment levels of additional growth factors that may be co- or counter- regulated with VEGF and correlate with response to treatment.
Time Frame: 1 year
Population: We initially planned to measure baseline and on treatment levels of coagulation and endothelial cell activation markers that may predict for thrombotic or bleeding risks related to treatment. These markers are best analyzed in citrated plasma and funding was not available for tube collection and analysis.
Arm/Group | BIBF 1120
Number analyzed (Participants) | 0

8. Other Pre Specified Outcome: VEGF Levels Correlated With Treatment Outcome
Description: Baseline levels of VEGF were correlated with treatment outcome. Results are stratified in groups: "Partial Response (PR) or Stable Disease (SD)" and "Progressive Disease (PD)"
Time Frame: 1 year
Population: VEGF levels measured and stratified into two groups: those who experienced either Partial Response (PR) or Stable Disease (SD); and those who experienced Progressive Disease (PD). Data was not collected for one subject
Measure: Median (Inter-Quartile Range); unit: picograms per milliliter
Arm/Group | BIBF 1120
Number analyzed (Participants) | 26
picograms per milliliter
  Partial Response or Stable Disease: number analyzed (Participants) | 11
  Partial Response or Stable Disease | 1405 [958 to 1580]
  Progressive Disease: number analyzed (Participants) | 15
  Progressive Disease | 1033 [698 to 1199]

9. Other Pre Specified Outcome: Concentration of Select Growth Factors Measured in Nanograms Per Milliliter Reported as a Function of Treatment Response
Description: Correlating baseline and on treatment levels of additional growth factors measured in nanograms per milliliter that may be co- or counter- regulated with VEGF with response to treatment
Time Frame: 1 year
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: nanograms per milliliter
Arm/Group | BIBF 1120
Number analyzed (Participants) | 26
nanograms per milliliter
  ICAM-1: Partial Response or Stable Disease: number analyzed (Participants) | 11
  ICAM-1: Partial Response or Stable Disease | 635.1 [584.0 to 688.0]
  ICAM-1: Progressive Disease: number analyzed (Participants) | 15
  ICAM-1: Progressive Disease | 686.8 [589.0 to 951.0]
  OPN: Partial Response or Stable Disease: number analyzed (Participants) | 11
  OPN: Partial Response or Stable Disease | 643.0 [470.0 to 887.0]
  OPN: Progressive Disease: number analyzed (Participants) | 15
  OPN: Progressive Disease | 923.0 [530.0 to 1349.0]
  TGF-Beta1: Partial Response or Stable Disease: number analyzed (Participants) | 11
  TGF-Beta1: Partial Response or Stable Disease | 122.5 [93.4 to 134.6]
  TGF-Beta1: Progressive Disease: number analyzed (Participants) | 15
  TGF-Beta1: Progressive Disease | 90.3 [75.8 to 118.4]
  TGF-Beta2: Partial Response or Stable Disease: number analyzed (Participants) | 11
  TGF-Beta2: Partial Response or Stable Disease | 22.0 [14.4 to 34.9]
  TGF-Beta2: Progressive Disease: number analyzed (Participants) | 15
  TGF-Beta2: Progressive Disease | 33.4 [14.4 to 57.2]
  TIMP-1: Partial Response or Stable Disease: number analyzed (Participants) | 11
  TIMP-1: Partial Response or Stable Disease | 93.5 [72.2 to 108.7]
  TIMP-1: Progressive Disease: number analyzed (Participants) | 15
  TIMP-1: Progressive Disease | 116.4 [88.2 to 141.9]
  TSP-2: Partial Response or Stable Disease: number analyzed (Participants) | 11
  TSP-2: Partial Response or Stable Disease | 95.1 [77.6 to 113.7]
  TSP-2: Progressive Disease: number analyzed (Participants) | 15
  TSP-2: Progressive Disease | 104.9 [91.5 to 169.4]

10. Other Pre Specified Outcome: Concentration of VCAM-1 Reported as a Function of Treatment Response
Description: Correlating baseline and on treatment levels of VCAM-1 measured in micrograms per milliliter that may be co- or counter- regulated with VEGF with response to treatment
Time Frame: 1 year
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: micrograms per milliliter
Arm/Group | BIBF 1120
Number analyzed (Participants) | 26
micrograms per milliliter
  VCAM-1: Partial Response or Stable Disease: number analyzed (Participants) | 11
  VCAM-1: Partial Response or Stable Disease | 2.2 [1.8 to 2.5]
  VCAM-1: Progressive Disease: number analyzed (Participants) | 15
  VCAM-1: Progressive Disease | 2.3 [1.6 to 2.8]

ADVERSE EVENTS:
Time Frame: The study period during which all AEs and SAEs are collected began after informed consent is obtained and initiation of study treatment on Cycle 1, Day 1. It ended 30 days following the last administration of study treatment, or if the patient initiated treatment with a new anti-cancer therapy, or study discontinuation/termination; whichever was earlier.
Arm/Group | BIBF 1120
All-Cause Mortality (participants affected / at risk) | 22/27
Serious Adverse Events (participants affected / at risk) | 6/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIBF 1120 (N=27)
Abdominal Pain (Gastrointestinal disorders) | 1
Kidney Infection (Infections and infestations) | 1
Non-cardiac chest pain (General disorders) | 1
Aspartate aminotransferase increased (Investigations) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BIBF 1120 (N=27)
Anemia (Blood and lymphatic system disorders) | 5
Leukocytosis (Blood and lymphatic system disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1 — Cold intolerance
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 9
Ascites (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 18
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 13
Chills (General disorders) | 1
Edema limbs (General disorders) | 5
Fatigue (General disorders) | 15
Fever (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 3
Infections and infestations - Other, specify (Infections and infestations) | 2 — One event: Ear infection One event: Fever blisters
Tooth infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 9
Alkaline phosphatase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 9
Creatinine increased (Investigations) | 3
Investigations - Other, specify (Investigations) | 1 — Alanine transaminase
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 3
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hyponatremia (Metabolism and nutrition disorders) | 5
Aarthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder- Other, specify (Musculoskeletal and connective tissue disorders) | 3 — One event: Ganglion cyst One event: Intermittent leg cramps One event: Arthralgia
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 9
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Bilateraly neuropathy, hands and feet
Peripheral sensory neuropathy (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Hematuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 4
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 — One event: Pelvic prolapse
Urinary frequency (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Vaginal pain (Reproductive system and breast disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 7
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/98/NCT01669798/Prot_SAP_000.pdf